CLINICAL TRIAL: NCT03620656
Title: FLASH-AF: The Validation of the FibriCheck Application for the Detection of Atrial Fibrillation
Brief Title: The Validation of the FibriCheck Application for the Detection of Atrial Fibrillation
Acronym: FLASH-AF
Status: Completed | Type: Observational
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; FibriCheck; Validation; Smartphone; Smartwatch
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The smartphone group: Patients recruited from the cardiology ward where 10 different smartphone devices will be used for the recording of PPG signals with the FibriCheck application. These recordings will be compared with single-lead ECG recorded with an AliveCor Smartphone devices and gold-standard 12-lead ECG to determine the diagnostic accuracy.
  Interventions: Diagnostic Test: FibriCheck
- The smartwatch group: Patients recruited from the cardiology ward where 2 different wearable devices will be used for the recording of PPG signals with the FibriCheck application. These recordings will be compared with single-lead ECG recorded with an AliveCor wearable and gold-standard 12-lead ECG to determine the diagnostic accuracy.
  Interventions: Diagnostic Test: FibriCheck

INTERVENTIONS:
Diagnostic Test: FibriCheck — Photoplethysmography-based smartphone or smartwatch sensor to assess cardiac rhythm

SUMMARY:
Optical sensing technologies have the potential to enable long-term heart rhythm monitoring. The medically certified and clinically validated FibriCheck technology has proven its value for spot-check measurements to detect AF. However, further validation and verification of this technology is necessary to evaluate the performance of the FibriCheck technology on different tools (smartphones and smartwatches). During this study the performance of various optical sensors, ranging from the camera in smartphones to the photodetector in smartwatches, will be explored and device and form-factor variability will be investigated. The objective is to define the accuracy of optical sensing systems in the detection of atrial fibrillation versus a reference traditional 12-lead ECG signal.

DETAILED DESCRIPTION:
During this study the performance of various optical sensors, ranging from the camera in smartphones to the photodetector in smartwatches, will be explored and device and form-factor variability will be investigated. The objective is to define the accuracy of optical sensing systems in the detection of atrial fibrillation versus a reference traditional 12-lead ECG signal. Therefore, 2 groups will be created where different technologies will be investigated i.e. Group 1 will use various mobile devices and Group 2 will use various wearable devices. The recruitment of patients will be carried out in the framework of the usual care practice, where patients can be recruited at different moments throughout their current care-cycle.

Group 1: Smartphone based sensor: Here, the user needs to place the finger on the smartphone camera for 60 seconds to obtain high quality PPG waveforms. These waveforms are analysed using automated algorithms and stored under a unique anonymized study ID.

Group 2: Smartwatch based sensor: Here, a wearable device is used that is placed on the wrist and will record a PPG signal, similar as the smartphone camera, but with a specific PPG sensor. The data is extracted and processed by the FibriCheck software and the algorithms generate a diagnostic output which is stored under a unique anonymized study ID.

The hardware involved originates from different providers. Since FibriCheck is certified as stand-alone software, it is expected that it functions independently from different hardware sources. This hypothesis will be addressed in this study.

Smartphone devices that will be used in this research: Samsung, Huawei, Xiaomi, Apple, LGE, Lenovo and ZTE devices. Wearable devices that will be used in this research: Apple and Fitbit smartwatch devices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* Pacemaker dependent heart rhythm
* Tremor or Parkinson's disease
* Barriers for communication and lack of capability to execute the handlings required for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without atrial fibrillation (based on 12-lead ECG) presenting at the cardiology ward for standard consultations or admitted for observation or cardiac interventions will be recruited.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy to identify atrial fibrillation | July 2019
  Assessment of the diagnostic accuracy of the FibriCheck smartphone or smartwatch application to detect atrial fibrillation on devices with various technical aspects. The diagnostic accuracy will be determined by comparing the FibriCheck diagnosis with the diagnosis of a gold-standard 12-lead ECG. Differences in diagnostic accuracy of FibriCheck on different hardware devices will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Grieten, PhD, Study Director — CEO
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided